CLINICAL TRIAL: NCT03256773
Title: Imaging of Human Epithelial Airway Using a High Resolution Micro OCT Catheter (Functional Anatomic Imaging of CF Patients With Early Lung Disease Using Micro OCT)
Brief Title: High Resolution Micro OCT Imaging
Status: Active, not recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Massachusetts General Hospital (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Steven M Rowe, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: F160125001; 1R01HL116213 (NIH)
Record Dates: First submitted 2017-08-18; First posted 2017-08-22 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Cystic Fibrosis; COPD; PCD - Primary Ciliary Dyskinesia; Covid19; Sinusitis
MeSH Terms: conditions — Cystic Fibrosis; Pulmonary Disease, Chronic Obstructive; Ciliary Motility Disorders; COVID-19; Sinusitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Notmal: No lung Disease
- Cystic Fibrosis: cystic fibrosis Lung Disease
- PCD: Primary Ciliary Dyskinesia
- COPD: Chronic Obstructive Lung Disease

SUMMARY:
The purpose of this study is to learn about using the imaging to make images of the lungs and nose with the long-term goal of the research leading to potential treatments and new therapies for patients with cystic fibrosis.

DETAILED DESCRIPTION:
Lung Disease is the predominate cause of morbidity and mortality in patients with cystic fibrosis (CF). A better understanding of the primary pathogenesis of CF is essential in order to reveal the features that may lead to the onset of progressive lung disease. Discerning the nature of the CF defect could resolve longstanding controversy and result in a new therapeutic opportunity that may address pathophysiology. Recently the investigators have developed an innovative technology, termed 1-µm resolution optical coherence tomography (µOCT), which enables real-time cross-sectional microscopy of the functional epithelial surface of living airways.

ELIGIBILITY:
THE INCLUSION CRITERIA:

* Patients diagnosed with CF or healthy normal controls with no respiratory disease
* Patients must be over the age of 14
* Patient must be able to give informed consent

THE EXCLUSION CRITERIA:

* Patients with recent respiratory infection requiring antibiotics or corticosteroids in the last 4 weeks (excluding routine perioperative antibiotics)
* Patients with major sinus surgery that will alter the nasal anatomy and preclude imaging of the nares
* Any condition that in the opinion of the investigator will alter the safety of pilot testing in the operating room
* Female subjects who are pregnant

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with CF, COPD, Sinusitis, PCD and COVID 19 will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-04-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
feasibility of uOCT probe | 1 year
  to determine if a uOCT probe can image airway epithelial cells from the lung and the nares of adult patients

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Rowe, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No